CLINICAL TRIAL: NCT00270296
Title: Lopinavir/Ritonavir/Combivir vs. Abacavir/Zidovudine/Lamivudine for Virologic Efficacy and the Prevention of Mother-to-Child HIV Transmission Among Breastfeeding Women With CD4 Counts Greater Than or Equal to 200 Cells/mm3 in Botswana
Brief Title: Trizivir Vs. Kaletra and Combivir for the Prevention of Mother-to-Child Transmission of HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BHP 016; U01AI064002 (NIH)
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Treatment Naive; MTCT; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — abacavir, lamivudine, and zidovudine drug combination; lamivudine, zidovudine drug combination; Lopinavir; Nevirapine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes

ARMS (3):
- Trizivir (TZV) Arm (Experimental): Participants in the TZV Arm (Arm 1A) will be pregnant women who have CD4 counts of 200 cells/mm3 or more. As the intervention, they will receive TZV twice daily. Once in labor, these participants will continue to take TZV twice daily and will also be given additional ZDV.
  Interventions: Drug: Trizivir
- Kaletra Arm (Experimental): Participants in the Kaletra Arm (Arm 1B) will be pregnant women who have CD4 counts of 200 cells/mm3 or more. As the intervention, they will receive Lamivudine/Zidovudine (3TC/ZDV) and Lopinavir/Ritonavir (LPV/RTV) twice daily. Once in labor, these participants will continue to take TZV twice daily and will also be given additional ZDV.
  Interventions: Drug: Lamivudine/Zidovudine; Drug: Lopinavir/Ritonavir
- Nevirapine (NVP) Arm (Experimental): Participants in the NVP Arm (Arm 2) will be pregnant women who have have CD4 counts less than 200 cells/mm3. These participants will receive NVP once daily for the first 14 days, then twice daily, and 3TC/ZDV twice daily; these women will be in the observational group.
  Interventions: Drug: Nevirapine

INTERVENTIONS:
Drug: Trizivir — 300 mg abacavir sulfate/150 mg lamivudine/300 mg zidovudine tablet taken orally twice daily
  Other Names: TZV
  Arms: Trizivir (TZV) Arm
Drug: Lamivudine/Zidovudine — 150 mg lamivudine/300 mg zidovudine tablet taken orally twice daily
  Other Names: 3TC/ZDV; Combivir
  Arms: Kaletra Arm
Drug: Lopinavir/Ritonavir — 400 mg lopinavir/100 mg ritonavir tablet taken orally twice daily
  Other Names: LPV/RTV
  Arms: Kaletra Arm
Drug: Nevirapine — 200 mg tablet taken orally daily for the first 14 days before receiving 200 mg tablet taken orally twice daily
  Other Names: NVP
  Arms: Nevirapine (NVP) Arm

SUMMARY:
Anti-HIV drug regimens have dramatically improved the rates of prevention of mother-to-child transmission (MTCT) of HIV in developed countries. However, little is known of the effectiveness of such regimens in developing countries, such as Botswana. This study will determine whether Trizivir (TZV), a single pill containing abacavir sulfate, lamivudine, and zidovudine (ABC/3TC/ZDV), or lopinavir/ritonavir (LPV/r) and lamivudine/zidovudine (3TC/ZDV) is more effective in reducing HIV-1 viral load and preventing MTCT among HIV infected pregnant women in Botswana.

DETAILED DESCRIPTION:
While perinatal HIV infection has become rare in developed countries through the use of highly active antiretroviral therapy (HAART), it remains a serious problem in developing countries. Botswana has a population of approximately 1.7 million; the prevalence of HIV in Botswana is about 37.4%. In the developed world, HAART has revolutionized the prevention of MTCT among nonbreastfed infants. This trial will compare the effectiveness of a protease inhibitor (PI)-based regimen versus a triple nucleoside reverse transcriptase inhibitor (NRTI)-based regimen in preventing MTCT of HIV.

This study will last up to 24 months for mothers and their children. Participants will be stratified based on their CD4 count at screening. Women with CD4 counts of 200 cells/mm3 or more will be in one of two treatment groups and will be randomly assigned to receive either TZV twice daily or LPV/RTV and 3TC/ZDV twice daily. Once in labor, treatment group participants will continue to take their assigned HAART regimen and will also be given additional ZDV. Women with CD4 counts less than 200 cells/mm3 will receive nevirapine (NVP) once daily for the first 14 days, then twice daily, and 3TC/ZDV twice daily; these women will be in the observational group.

Shortly after birth, infants will receive single-dose NVP. A 1-month supply of ZDV will be provided to the mother to administer daily to her child. Mothers will stop HAART at 6 months postpartum or when they stop breastfeeding, whichever occurs earlier. A clinical evaluation, blood collection, and HIV prevention counseling will occur at all maternal visits. An obstetrical exam and physical exam will occur at selected visits. Women will provide at least four samples of breast milk during the first 5 months postpartum. For infants, a clinical evaluation will occur at every visit, and a physical exam and blood collection will occur at selected visits.

ELIGIBILITY:
Inclusion Criteria for Mothers:

* HIV-infected
* At least at 26th week of pregnancy (treatment group) or 18th week of pregnancy (observational group) but not beyond the 34th week of pregnancy
* Able to complete study visits until at least 6 months postpartum
* Citizen of Botswana

Exclusion Criteria for Mothers:

* Taken ARVs for more than 1 week, other than ZDV, during current or prior pregnancy. Women who have received single-dose NVP in a prior pregnancy are not excluded.
* Certain abnormal laboratory values
* Plan to formula feed
* Known fetal abnormalities that suggest the fetus will not survive to 6 months of gestational age
* Known allergy or medical contraindication to any of the study drugs
* Require certain medications
* Previous participation in the "Prevention of Milk-Borne Transmission of HIV-1C in Botswana" (Mashi) study
* Currently incarcerated

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Shapiro, MD, MPH, Principal Investigator — Division of Infectious Diseases, Beth Israel Deaconess Medical Center, Botswana-Harvard School of Public Health Partnership for Research and Education; Claire Moffat, MD, MPH, Principal Investigator — Department of Immunology and Infectious Diseases, Harvard School of Public Health, Botswana-Harvard School of Public Health Partnership for Research and Education
Locations (4):
- Botswana (4):
  - Princess Marina Hosp., BHP Study Clinic, Gaborone Shapiro CRS, Gaborone
  - Athlone Hosp., BHP Study Clinic, Lobatse Shapiro CRS, Lobatse
  - Deborah Reteif Hosp., BHP Study Clinic, Mochudi Shapiro CRS, Mochudi
  - Scottish Livingstone Hosp., BHP Study Clinic, Molepolole Shapiro CRS, Molepolole

REFERENCES:
- [Background] Cooper ER, Charurat M, Mofenson L, Hanson IC, Pitt J, Diaz C, Hayani K, Handelsman E, Smeriglio V, Hoff R, Blattner W; Women and Infants' Transmission Study Group. Combination antiretroviral strategies for the treatment of pregnant HIV-1-infected women and prevention of perinatal HIV-1 transmission. J Acquir Immune Defic Syndr. 2002 Apr 15;29(5):484-94. doi: 10.1097/00126334-200204150-00009. PMID 11981365
- [Background] Dorenbaum A, Cunningham CK, Gelber RD, Culnane M, Mofenson L, Britto P, Rekacewicz C, Newell ML, Delfraissy JF, Cunningham-Schrader B, Mirochnick M, Sullivan JL; International PACTG 316 Team. Two-dose intrapartum/newborn nevirapine and standard antiretroviral therapy to reduce perinatal HIV transmission: a randomized trial. JAMA. 2002 Jul 10;288(2):189-98. doi: 10.1001/jama.288.2.189. PMID 12095383
- [Background] Jones BM, Chiu SS, Wong WH, Lim WW, Lau YL. Cytokine profiles in human immunodeficiency virus-infected children treated with highly active antiretroviral therapy. MedGenMed. 2005 May 3;7(2):71. PMID 16369449
- [Background] Moodley D, Moodley J, Coovadia H, Gray G, McIntyre J, Hofmyer J, Nikodem C, Hall D, Gigliotti M, Robinson P, Boshoff L, Sullivan JL; South African Intrapartum Nevirapine Trial (SAINT) Investigators. A multicenter randomized controlled trial of nevirapine versus a combination of zidovudine and lamivudine to reduce intrapartum and early postpartum mother-to-child transmission of human immunodeficiency virus type 1. J Infect Dis. 2003 Mar 1;187(5):725-35. doi: 10.1086/367898. Epub 2003 Feb 24. PMID 12599045
- [Background] Richardson BA, John-Stewart GC, Hughes JP, Nduati R, Mbori-Ngacha D, Overbaugh J, Kreiss JK. Breast-milk infectivity in human immunodeficiency virus type 1-infected mothers. J Infect Dis. 2003 Mar 1;187(5):736-40. doi: 10.1086/374272. Epub 2003 Feb 12. PMID 12599046
- [Background] Rousseau CM, Nduati RW, Richardson BA, Steele MS, John-Stewart GC, Mbori-Ngacha DA, Kreiss JK, Overbaugh J. Longitudinal analysis of human immunodeficiency virus type 1 RNA in breast milk and of its relationship to infant infection and maternal disease. J Infect Dis. 2003 Mar 1;187(5):741-7. doi: 10.1086/374273. Epub 2003 Feb 18. PMID 12599047
- [Derived] Powis KM, Smeaton L, Hughes MD, Tumbare EA, Souda S, Jao J, Wirth KE, Makhema J, Lockman S, Fawzi W, Essex M, Shapiro RL. In-utero triple antiretroviral exposure associated with decreased growth among HIV-exposed uninfected infants in Botswana. AIDS. 2016 Jan;30(2):211-20. doi: 10.1097/QAD.0000000000000895. PMID 26684818
- [Derived] Powis K, Lockman S, Smeaton L, Hughes MD, Fawzi W, Ogwu A, Moyo S, van Widenfelt E, von Oettingen J, Makhema J, Essex M, Shapiro RL. Vitamin D insufficiency in HIV-infected pregnant women receiving antiretroviral therapy is not associated with morbidity, mortality or growth impairment in their uninfected infants in Botswana. Pediatr Infect Dis J. 2014 Nov;33(11):1141-7. doi: 10.1097/INF.0000000000000428. PMID 25037041
- [Derived] Shapiro RL, Kitch D, Ogwu A, Hughes MD, Lockman S, Powis K, Souda S, Moffat C, Moyo S, McIntosh K, van Widenfelt E, Zwerski S, Mazhani L, Makhema J, Essex M. HIV transmission and 24-month survival in a randomized trial of HAART to prevent MTCT during pregnancy and breastfeeding in Botswana. AIDS. 2013 Jul 31;27(12):1911-20. doi: 10.1097/qad.0b013e32836158b0. PMID 24180000
- [Derived] Dryden-Peterson S, Jayeoba O, Hughes MD, Jibril H, McIntosh K, Modise TA, Asmelash A, Powis KM, Essex M, Shapiro RL, Lockman S. Cotrimoxazole prophylaxis and risk of severe anemia or severe neutropenia in HAART-exposed, HIV-uninfected infants. PLoS One. 2013 Sep 23;8(9):e74171. doi: 10.1371/journal.pone.0074171. eCollection 2013. PMID 24086319
- [Derived] Dryden-Peterson S, Shapiro RL, Hughes MD, Powis K, Ogwu A, Moffat C, Moyo S, Makhema J, Essex M, Lockman S. Increased risk of severe infant anemia after exposure to maternal HAART, Botswana. J Acquir Immune Defic Syndr. 2011 Apr 15;56(5):428-36. doi: 10.1097/QAI.0b013e31820bd2b6. PMID 21266910
- [Derived] Powis KM, Smeaton L, Ogwu A, Lockman S, Dryden-Peterson S, van Widenfelt E, Leidner J, Makhema J, Essex M, Shapiro RL. Effects of in utero antiretroviral exposure on longitudinal growth of HIV-exposed uninfected infants in Botswana. J Acquir Immune Defic Syndr. 2011 Feb 1;56(2):131-8. doi: 10.1097/QAI.0b013e3181ffa4f5. PMID 21124227
- [Derived] Shapiro RL, Hughes MD, Ogwu A, Kitch D, Lockman S, Moffat C, Makhema J, Moyo S, Thior I, McIntosh K, van Widenfelt E, Leidner J, Powis K, Asmelash A, Tumbare E, Zwerski S, Sharma U, Handelsman E, Mburu K, Jayeoba O, Moko E, Souda S, Lubega E, Akhtar M, Wester C, Tuomola R, Snowden W, Martinez-Tristani M, Mazhani L, Essex M. Antiretroviral regimens in pregnancy and breast-feeding in Botswana. N Engl J Med. 2010 Jun 17;362(24):2282-94. doi: 10.1056/NEJMoa0907736. PMID 20554983

RESULTS

PARTICIPANT FLOW:
Groups:
- TZV Arm: Participants in Arm 1A will have CD4 counts of 200 cells/mm3 or more and will receive TZV twice daily. Once in labor, these participants will continue to take TZV twice daily and will also be given additional ZDV.
  Trizivir: 300 mg abacavir sulfate/150 mg lamivudine/300 mg zidovudine tablet taken orally twice daily
- Kaletra Arm: Participants in Arm 1B will have CD4 counts of 200 cells/mm3 or more and will receive LPV/RTV and 3TC/ZDV twice daily. Once in labor, these participants will continue to take TZV twice daily and will also be given additional ZDV.
  Lamivudine/Zidovudine: 150 mg lamivudine/300 mg zidovudine tablet taken orally twice daily
  Lopinavir/Ritonavir: 400 mg lopinavir/100 mg ritonavir tablet taken orally twice daily
- NVP Arm: Participants in Arm 2 will have CD4 counts less than 200 cells/mm3 and will receive NVP once daily for the first 14 days, then twice daily, and 3TC/ZDV twice daily; these women will be in the observational group.
  Nevirapine: 200 mg tablet taken orally daily for the first 14 days before receiving 200 mg tablet taken orally twice daily
Period: Overall Study
Arm/Group | TZV Arm | Kaletra Arm | NVP Arm
Started | 285 | 275 | 170
Completed | 186 | 185 | 109
Not Completed | 99 | 90 | 61

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TZV Arm | Kaletra Arm | NVP Arm | Total
Number analyzed (Participants) | 285 | 275 | 170 | 730
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 285 | 275 | 170 | 730
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 275 | 170 | 730
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 285 | 275 | 170 | 730
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Botswana | 285 | 275 | 170 | 730

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Virologic Suppression
Description: Suppression of the plasma HIV-1 RNA level to less than 400 copies per milliliter
Time Frame: Throughout study, including breastfeeding, assessed up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | TZV Arm | Kaletra Arm | NVP Arm
Number analyzed (Participants) | 285 | 275 | 170
Participants | 274 | 256 | 160

2. Primary Outcome: Number of HIV+ Infants
Description: Number of infants with HIV-positive status
Time Frame: Throughout study, including breastfeeding, assessed up to 24 months
Population: Analysis is based on actual number of available patients, and may not perfectly match the Patient Flow module.
Measure: Number; unit: Infants
Arm/Group | TZV Arm | Kaletra Arm | NVP Arm
Number analyzed (Participants) | 283 | 270 | 156
Infants | 6 | 1 | 1

ADVERSE EVENTS:
Arm/Group | TZV Arm | Kaletra Arm | NVP Arm
All-Cause Mortality (participants affected / at risk) | 1/285 | 0/275 | 3/170
Serious Adverse Events (participants affected / at risk) | 42/285 | 32/275 | 48/170
Other Adverse Events (participants affected / at risk) | 0/285 | 0/275 | 0/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TZV Arm (N=285) | Kaletra Arm (N=275) | NVP Arm (N=170)
Grade 3 or 4 Laboratory Event (Blood and lymphatic system disorders) | 42 | 32 | 48 — Neutropenia or anemia or liver function test (LFT) abnormality

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No